CLINICAL TRIAL: NCT04593199
Title: Physical Activity Promotion in Children Using a Novel Smartphone Game: A Pilot Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Sam Liu, Assistant Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UVic181243
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Physical Activity
Keywords: Children; Mobile health; Gamification; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Tracking App Only (Sham Comparator): Over a four week period, participants were asked to use the Fitbit app to track their daily physical activity.
  Interventions: Behavioral: Physical activity tracking app
- Physical Activity Tracking + Gamified Smartphone App (Active Comparator): Over a four week period, participants were asked to use the Fitbit app to track their daily physical activity. Additionally, they were asked to use the gamified smartphone app, Draco, during the intervention period.
  Interventions: Behavioral: Gamified Smartphone App

INTERVENTIONS:
Behavioral: Gamified Smartphone App — The primary objective was to determine the acceptability and satisfaction of the Draco app among children. Secondary objective was to evaluate if the Draco app could improve physical activity levels (steps, and moderate-to-vigorous physical activity) and intrinsic motivation for physical activity in children. The gamified smartphone app, Draco, is a virtual pet simulator where you care for a pet by exercising, walking, and answering healthy lifestyle questions.
  Other Names: Draco app
  Arms: Physical Activity Tracking + Gamified Smartphone App
Behavioral: Physical activity tracking app — Participants were asked to use the Fitbit app to track and sync their daily physical activity.
  Other Names: Fitbit app
  Arms: Physical Activity Tracking App Only

SUMMARY:
Increasing physical activity is critical for children's overall health. Smartphone apps using gamification has shown promise to increasing physical activity using game techniques. This study is a 4-week randomized controlled trial using a gamified smartphone app to determine acceptability and preliminary effectiveness to increase physical activity in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-14 years old
* Not meeting the recommended Canadian physical activity guidelines of 60min per day of moderate-to-vigorous physical activity
* English-literate
* Normal to corrected vision

Exclusion Criteria:

* Diagnosis or injury that prevents physical activity participation
* No access to a smartphone or tablet

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
User satisfaction with gamified smartphone app | 4 weeks
  User satisfaction was measured using an adapted version of the short form Intrinsic Motivation Inventory used by Ahn, Johnsen & Ball, 2019. Items pertained to the enjoyment, satisfaction of using the app and if the experience was unenjoyable. Scores are rated on a 5 point Likert scale where 1 is the lowest score and 5 is the highest. 1 = Not true for me; 2 = Not really true for me; 3 = Sometimes true for me; 4 = Often true for me; 5 = Very true for me.
Acceptability with gamified smartphone app | 4 weeks
  Exit interviews were performed after the intervention period to determine satisfaction and acceptability. Questions related to their experience using the app, their physical activity behavior (before, during, and after the intervention period) and recommendations for app content

SECONDARY OUTCOMES:
Steps | 4 weeks
  Steps were collected using a Fitbit over the intervention period. Fitbit is a previously validated and reliable instrument to measure physical activity (Feehan et al., 2018).
Physical activity minutes | 4 weeks
  Minutes of physical activity engaged in by the participants were collected using a Fitbit device worn by participants. The device is worn while the participant is engaging in physical activity. The intensity of exercise is calculated by heartrate. Fitbit is a previously validated and reliable instrument to measure physical activity (Feehan et al., 2018).
Motivation for physical activity | 4 weeks
  Motivation for physical activity was measured using an adapted version of the Intrinsic Motivation Inventory used by Ahn, Johnsen & Ball, 2019. Questions related to perceived competence to physical activity, perceived autonomy to physical activity and perceived relatedness to the app. The items addressed perceived competence, perceived autonomy, and relatedness. Scores are rated on a 5 point Likert scale where 1 is the lowest score and 5 is the highest. 1 = Not true for me; 2 = Not really true for me; 3 = Sometimes true for me; 4 = Often true for me; 5 = Very true for me.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided